CLINICAL TRIAL: NCT03942276
Title: Acute and Chronic Health Effects of Different Exercises Interventions in Post-menopausal Women: a Clinical, Controlled and Randomized Study
Brief Title: Effects of Different Exercises Interventions in Post-menopausal Women
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Participants constantly reported knee pain.
Sponsor: Federal University of Uberlandia (Other)
Responsible Party: Principal Investigator, Igor Moraes Mariano, Principal investigator, Federal University of Uberlandia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CEP UFU 07839218.8.0000.5152
Record Dates: First submitted 2019-04-24; First posted 2019-05-08 (Actual); Last update posted 2021-01-11 (Actual); Status verified 2021-01

CONDITIONS: Hypertension; Menopause
Keywords: Blood pressure; Menopause; Hypertension; Exercise; Alternative training
MeSH Terms: conditions — Hypertension; Motor Activity | interventions — High-Intensity Interval Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Placebo Comparator): Hypertensive post menopausal women, who will do the evaluations before the beginning and after 12 weeks without perform exercise training.
  Interventions: Other: Control
- Alternative training (Experimental): Hypertensive post menopausal women, who will do the evaluations before the beginning and after 12 weeks of high intensity interval training.
  Interventions: Other: High intensity interval training
- Conventional training (Experimental): Hypertensive post menopausal women, who will do the evaluations before the beginning and after 12 weeks of moderate intensity continuous training
  Interventions: Other: Moderate intensity continuous training

INTERVENTIONS:
Other: High intensity interval training — Consists of 60 seconds sets of high-intensity exercises, characterized by heart rate> 85% of maximal heart rate (HRmax), obtained through the formula (220-age), or by the Rated Perceived Exertion between 7 and 8 on the Borg scale, which ranges from 0 to 10. Of the 60 seconds of high intensity exercise, 30 seconds will be to get up and down a 16 cm step and 30 seconds of squats, with knee flexion greater than 90º, both at the highest possible speed. The recovery between sets is light walk for 60 seconds. If the volunteers do not reach the proposed intensity zone, they will be instructed to increase the number of squats and step ascents and descents.
  Other Names: Alternative aerobic exercise training
  Arms: Alternative training
Other: Moderate intensity continuous training — Consist of performing a 30 minute walk at 50% of reserve heart rate (HRR), calculated by (HRmax - HRmax) x% + HRmax. HRmax being obtained by means of the formula (220 - age).
  Other Names: Traditional aerobic exercise training
  Arms: Conventional training
Other: Control — Consist of performing no exercise training.
  Arms: Control

SUMMARY:
This study will compare different exercise training protocols on health parameters of postmenopausal women. The hypothesis is that short duration high intensity interval training will promote different effects of long duration moderate intensity training.

DETAILED DESCRIPTION:
Exercise load control still not a consensus as to the most effective strategy for improving health parameters in postmenopausal women. In this way, the volunteers will perform anthropometric and body composition assessments, climacteric symptoms and sleep quality evaluations, blood pressure reactivity, resting blood pressure and heart rate and ambulatorial blood pressure monitoring, before and after 12 weeks of training.

ELIGIBILITY:
Inclusion Criteria:

* being postmenopausal (amenorrhea of at least 12 months and [FSH]> 40 mlU/ml); be controlled hypertension; not to undergo drug treatment with β-blockers; not make use of sex hormone therapies; do not present physical problems or cardiovascular complications that prevent the performance of physical exercises; present attestation of a cardiologist proving that they are able to perform physical exercises.

Exclusion Criteria:

* Do not attend the collection site on the day and time programmed more than once in the acute phase of the study; missing more than 2 consecutive sessions or 6 alternates in the chronic phase of the study; unable to perform the proposed training protocols; change in drug therapy during the intervention.

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Changes in Ambulatorial Blood Pressure | Before and within 72 hours after 12 weeks of exercise training/control
  All volunteers were submitted to a 24-hour Blood Pressure (BP) assessment by Ambulatorial Blood Pressure Monitoring (ABPM) before and after 10 weeks of combined exercise training, with a minimum of 48 hours after the last training session. A device was used associated with a diary of examination to self-report of activities of daily living (sleep, work, food) or any event that could interfere abnormally with BP or device measurements. The device was always placed 7am and the measurements were made every 15 minutes from 7h to 23h and every 30 minutes from 23h to 7h. The monitoring was considered valid when it happened for a period of 24 hours. The following results were evaluated: systolic blood pressure; diastolic blood pressure and mean blood pressure in awake, sleep and 24-hour periods, and shall be expressed in mmHg.
Changes in Resting Blood Pressure | Before and within 72 hours after 12 weeks of exercise training/control
  Before the use ABPM during daily activities, resting blood pressure were measured using the same equipment after 15 min of rest in siting position. The following results were evaluated: systolic blood pressure; diastolic blood pressure and mean blood pressure, they shall be expressed in mmHg.

SECONDARY OUTCOMES:
Changes in Heart Rate Variability | Before and within 72 hours after 12 weeks of exercise training/control
  Heart Rate (HR) was recorded using a heart rate monitor in a beat-by-beat basis. HR was registered in a seat position for 20 min of rest. Prior to the HR Variability (HRV) analysis, the RR intervals (RRi) were visually inspected and filtered using a moving average filter. The HRV was analyzed in both time-, frequency- and nonlinear-domain. Being that for frequency-domain analysis, firstly the RRi series were interpolated at 4 Hz and then the signal linear trend component removal was performed using the smooth priors approach.
Changes in Ambulatorial Blood Pressure Variability | Before and within 72 hours after 12 weeks of exercise training/control
  Based on Ambulatorial Blood Pressure data, were calculated Blood Pressure Variability by: 24-hour standard deviation weighted by the time interval between consecutive readings; the mean diurnal and nocturnal deviations weighted for the duration of the daytime and nighttime interval; the average real variability weighted for the time interval between consecutive readings; the ambulatory arterial stiffness index calculated by the slope of the trend curve of the dispersion of pressure data; the morning surge that represents the dynamic daytime variation in morning pressure that tends to increase, being assessed from the point of least pressure during sleep in relation to the first two hours after waking; and nocturnal dipping, that represents the average percentage drop of sleep pressure in relation to wakefulness, and individuals with falls of 10% or more are considered dippers and below that are considered nom-dippers.
Changes in Blood pressure reactivity | Before and within 72 hours after 12 weeks of exercise training/control
  To evaluate blood pressure reactivity under mental stress, it will be used the 3 minutes Stroop protocol of words and colors. The test consists of a video on a computer screen facing the volunteer that changes the image every 2 seconds. The volunteer should then speak as quickly as possible the color of the letters present on the screen, being that in each image there is dissonance between the background color, the color of the letters and the word formed (which is always the name of another color ). At the end of the test, the volunteer demonstrates on a scale her difficulty in the test, according to the following classification: 0 = not stressful; 1 = slightly stressful; 3 = very stressful; and 4 = extremely stressful. Each minute of the test the blood pressure will be measured by auscultatory method, with stethoscope and mercury column, and the following results were evaluated: systolic blood pressure and diastolic blood pressure.
Changes in salivary oxidative stress (umol/L) | Before and within 72 hours after 12 weeks of exercise training/control
  The salivary was collected after 12-hours fasting and the total antioxidant capacity was evaluated using the Ferric-Ability of Plasma (FRAP) methodology and calculated from the standard trolox curve and the Lipid peroxidation levels were determined by the TBARS method (thiobarbituric acid reactive substances), using as standard a curve of 1,1,3,3-tetraethoxypropane (TMP). The total protein concentration was obtained by the Bradford method, using bovine serum albumin (BSA) as standard. Expressed in umol/L. Expressed in umol/L.
Changes in salivary oxidative stress (units/mg prot) | Before and within 72 hours after 12 weeks of exercise training/control
  The salivary was collected after 12-hours fasting and the activity of the enzyme superoxide dismutase (SOD) was determined based on the auto oxidation capacity of pyrogallol. Expressed in Units/ mg prot.
Changes in salivary oxidative stress (μmol H2O2/min/g prot) | Before and within 72 hours after 12 weeks of exercise training/control
  The salivary was collected after 12-hours fasting and the catalase activity (CAT) was calculated by monitoring the consumption of hydrogen peroxide at 240 nm. Expressed in μmol H2O2/min/g prot.
Changes in salivary oxidative stress (nM) | Before and within 72 hours after 12 weeks of exercise training/control
  The salivary was collected after 12-hours fasting and the amounts of nitric oxide (NO) were estimated by the determination of total nitrite by the Griess colorimetric method. Expressed in nM.
Changes in blood biomarkers (mg/dL) | Before and within 72 hours after 12 weeks of exercise training/control
  Samples of fasting venous blood (12 hours) will be collected in a sterile environment, using disposable materials. After local asepsis, 15 mL of blood will be obtained. Blood samples will be deposited in test tubes containing EDTA and dried tubes with separator gel for collection of serum. The samples will then be centrifuged at 1500 rpm for 15 minutes to separate plasma and serum aliquots and stored at -80 ° C. Will be used commercial ELISA-specific kits In order to determine the activity of C-reactive protein (CRP), total cholesterol, triglycerides, HDL cholesterol (HDL-C), LDL cholesterol (LDL-C) and Tryglicerides, all express in mg/dL. VLDL will be calculated using the equation suggested by the Brazilian Society of Cardiology, dividing the concentration of triglycerides by 5.
Changes in blood biomarkers (nM) | Before and within 72 hours after 12 weeks of exercise training/control
  Samples of fasting venous blood (12 hours) will be collected in a sterile environment, using disposable materials. After local asepsis, 15 mL of blood will be obtained. Blood samples will be deposited in test tubes containing EDTA and dried tubes with separator gel for collection of serum. The samples will then be centrifuged at 1500 rpm for 15 minutes to separate plasma and serum aliquots and stored at -80 ° C. Will be used commercial ELISA-specific kits In order to determine the activity of nitrite (NO-2) and nitrate (NO-3), expressed in nM.
Changes in blood biomarkers (pg/mL) | Before and within 72 hours after 12 weeks of exercise training/control
  Samples of fasting venous blood (12 hours) will be collected in a sterile environment, using disposable materials. After local asepsis, 15 mL of blood will be obtained. Blood samples will be deposited in test tubes containing EDTA and dried tubes with separator gel for collection of serum. The samples will then be centrifuged at 1500 rpm for 15 minutes to separate plasma and serum aliquots and stored at -80 ° C. Will be used commercial ELISA-specific kits In order to determine the activity of Interleukin-6 (IL-6), Interleukin-10 (IL-10) and Tumor Necrosis Factor α (TNFα), expressed in pg/mL.
Changes in blood biomarkers (mg/L) | Before and within 72 hours after 12 weeks of exercise training/control
  Samples of fasting venous blood (12 hours) will be collected in a sterile environment, using disposable materials. After local asepsis, 15 mL of blood will be obtained. Blood samples will be deposited in test tubes containing EDTA and dried tubes with separator gel for collection of serum. The samples will then be centrifuged at 1500 rpm for 15 minutes to separate plasma and serum aliquots and stored at -80 ° C. Will be used commercial ELISA-specific kits In order to determine the activity of Adiponectin concentration, expressed in mg/L.
Changes in blood biomarkers (Units/mg de prot) | Before and within 72 hours after 12 weeks of exercise training/control
  Samples of fasting venous blood (12 hours) will be collected in a sterile environment, using disposable materials. After local asepsis, 15 mL of blood will be obtained. Blood samples will be deposited in test tubes containing EDTA and dried tubes with separator gel for collection of serum. The samples will then be centrifuged at 1500 rpm for 15 minutes to separate plasma and serum aliquots and stored at -80 ° C. Will be used commercial ELISA-specific kits In order to determine the activity of Superoxide Dismutase (SOD) and Catalase (CAT), expressed in Units/mg de prot.
Changes in blood biomarkers (umol/L) | Before and within 72 hours after 12 weeks of exercise training/control
  Samples of fasting venous blood (12 hours) will be collected in a sterile environment, using disposable materials. After local asepsis, 15 mL of blood will be obtained. Blood samples will be deposited in test tubes containing EDTA and dried tubes with separator gel for collection of serum. The samples will then be centrifuged at 1500 rpm for 15 minutes to separate plasma and serum aliquots and stored at -80 ° C. Will be used commercial ELISA-specific kits In order to determine the activity of Thiobarbituric Acid (TBARS), expressed in umol/L.

CONTACTS AND LOCATIONS:
Locations (1):
- Guilherme Morais Puga, Uberlândia, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: Undecided